CLINICAL TRIAL: NCT03796481
Title: Sleep, Pain and Function in People With Chronic Spinal Pain and Comorbid Insomnia Compared to People With Chronic Spinal Pain Without Insomnia.
Brief Title: Sleep, Pain and Function in People With Chronic Spinal Pain and Comorbid Insomnia
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Vrije Universiteit Brussel (Other); University Hospital, Ghent (Other); Universitair Ziekenhuis Brussel (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2018/0277/Amend
Record Dates: First submitted 2018-12-19; First posted 2019-01-08 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Chronic Low Back Pain; Chronic Neck Pain; Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: People with chronic spinal pain (i.e. chronic low back pain or chronic neck pain) with comorbid insomnia
- Controls: People with chronic spinal pain (i.e. chronic low back pain or chronic neck pain) without comorbid insomnia

SUMMARY:
This study is focused on people with chronic spinal pain. To investigate the impact of sleep problems on pain and function, 45 people with chronic spinal pain and comorbid insomnia will be compared to 45 people with chronic spinal pain without insomnia.

ELIGIBILITY:
Inclusion criteria cases:

* nonspecific spinal pain (≥3 days per week and ≥3 months of chronic low back pain, failed back surgery syndrome > 3 years prior, chronic whiplash, or chronic non traumatic neck pain)
* aged between 18 and 65 years
* seeking care because of neck pain or low back pain
* native dutch speaker
* having insomnia: in the absence of other intrinsic sleep disorders and shift work, insomnia is defined as > 30 minutes of sleep latency and/or minutes awake after sleep onset for > 3 days / week for > 6 months
* living or working within a radius of 50 km around the test location
* not starting new treatments or medication and continuing their usual care 6 weeks prior to and during study participation (to obtain steady state)
* referring from analgesics, caffeine, alcohol or nicotine in the previous 48 h of the assessments
* nonspecific failed back surgery > 3 years are permitted
* not undertaking exercise (>3 metabolic equivalents) 3 days before the experiment

Exclusion criteria cases:

* severe underlying sleep pathology (identified through baseline data of polysomnography)
* neuropathic pain
* chronic widespread pain
* being pregnant or pregnancy (including giving birth) in the preceding year
* history of specific spinal surgery
* thoracic pain in absence of neck or low back pain
* shift workers
* present clinical depression
* BMI ≥ 30

Inclusion criteria controls:

* native dutch speaking
* 18 to 65 years of age
* having chronic nonspecific chronic spinal pain (≥3 days per week and ≥3 months of chronic low back pain, failed back surgery syndrome > 3 years prior, chronic whiplash, or chronic non traumatic neck pain)
* referring from analgesics, caffeine, alcohol or nicotine in the previous 48 h of the assessments
* not undertaking exercise (>3 metabolic equivalents) 3 days before the experiment
* No new medication 6 weeks prior to the assessment
* currently not undergoing any treatment (excl. medication) for chronic spinal pain

Exclusion criteria controls:

* specific medical conditions (neuropathic pain, specific neck of back surgery, osteoporotic vertebral fractures, or rheumatologic diseases)
* chronic widespread pain syndromes (fibromyalgia or chronic fatigue syndrome)
* having insomnia (in the absence of other intrinsic sleep disorders and shift work, insomnia is defined as > 30 minutes of sleep latency and/or minutes awake after sleep onset for > 3 days / week for > 6 months)
* severe underlying sleep pathology
* being pregnant or pregnancy in the preceding year
* thoracic pain in the absence of neck or low back pain
* diagnosed depression
* BMI over 30

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with chronic spinal pain with and without comorbid insomnia (cases vs controls)
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (Numeric Rating Scale): Pain intensity | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported pain: The question "please rate your pain by circling the one number that best describes your pain on the AVERAGE" is used as the primary outcome measure to evaluate pain intensity. Scale ranges from 0 to 10, with higher scores indicating more self-reported pain.

SECONDARY OUTCOMES:
Brief Pain Inventory: Pain Interference | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported central sensitization symptoms. Score ranges from 0 to 100, with higher scores indicating more self-reported symptoms of central sensitization.
Central sensitization Inventory | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported central sensitization symptoms. Score ranges from 0 to 100, with higher scores indicating more self-reported symptoms of central sensitization.
Pressure Pain Thresholds | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Pressure Pain Thresholds at measured bilaterally with a digital pressure algometer (Wagner Instruments), both at symptomatic levels (trapezius muscle and 5 centimetres lateral to the spinous process of L3) and at remote sites (i.e. secondary hyperalgesia).
Sleep: Polysomnography (PSG) using the portable Alice PDX system, Philips Respironics Inc | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Participants will be monitored in the comfort of their own home by ambulatory polysomnography. This will provide the following parameters: time in bed, total sleep time, sleep onset latency, wake duration after sleep onset, early morning awakening, sleep staging, sleep efficiency, sleep fragmentation, respiratory parameters, cardiac and myoclonic activity.
Pittsburg Sleep Quality Index | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported perceived sleep quality. Score ranges from 0 to 21, 0 indicating no difficulty and 21 indicating severe sleep difficulties.
Insomnia Severity Index | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported insomnia severity. Score ranges from 0 to 28, with 0 indicating no clinically significant insomnia and 28 indicating severe clinical insomnia.
DBAS (i.e. Dysfunctional Beliefs and Attitudes about Sleep) | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Change in self-reported dysfunctional beliefs and attitudes about sleep. Score ranges from 0 to 10. Scores above 4 indicate unrealistic expectations for sleep or unrealistic thoughts about sleep.
Epworth Sleepiness Scale | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported sleep propensity. Score ranges from 0 to 24, with 0 indicating normal daytime sleepiness and 24 indicating severe excessive daytime sleepiness.
Brugmann Fatigue Scale | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported fatigue severity. Score ranges from 0 to 24, with higher scores indicating higher subjective levels of fatigue.
Hospital Anxiety and Depression rating scale | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported affective symptoms. Score ranges from 0 to 21, with 0 indicating absence of depression or anxiety and 21 indicating the presence of depression or anxiety.
Physical Activity using Actigraphy | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Physical activity: Continuous assessment of physical activity and rest/activity cycles
Short Form Health Survey - 36 items Mental Health | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported functional status and well-being or quality of life. Score ranges from 0 to 400 with higher scores indicating better mental health.
Short Form Health Survey - 36 items Physical Health | Participants will be tested one time only (one assessment) at one day, in between January 20, 2019 and April 30, 2021.
  Self-reported functional status and well-being or quality of life. Score ranges from 0 to 400 with higher scores indicating better physical health.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Vrije Universiteit Brussel, Brussels
  - Ghent University, Ghent